CLINICAL TRIAL: NCT06857071
Title: Site-randomized Trial of a Novel Social Network Recruitment Intervention to Locate More Undiagnosed Positive Cases of HIV, Increase HIV Testing Among Men, and Reduce HIV-related Stigma in South Africa (E-SNRHT South Africa)
Brief Title: Site-randomized Trial of an Expanded Social Network Recruitment to HIV Testing (E-SNRHT) Intervention to Locate Undiagnosed Cases and Reduce HIV-related Stigma
Acronym: E-SNRHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Human Sciences Research Council (Other Government); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH136871 (NIH); R01MH136871 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Undiagnosed HIV Infection; Populations That Are Reluctant to Test for HIV; Long-term Undiagnosed HIV Infection; Individuals With Newly-diagnosed HIV Infection; HIV-related Stigma; Access to HIV Testing
Keywords: expanded social network recruitment; social network recruitment to HIV testing; long-term undiagnosed HIV infection; HIV-related stigma; access to HIV testing; newly-diagnosed HIV infection; HIV testing intervention
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-SNRHT Intervention Arm (Experimental): The E-SNRHT intervention arm will recruit people newly diagnosed with HIV as "seeds" from clinics randomly assigned to the intervention condition, briefly remind them of HIV transmission risks and how HIV spreads through networks, and ask them to recruit people in their expanded social networks (i.e., anyone they know) who they think might benefit from being tested for HIV, whether or not they have engaged in any HIV risk behaviors together. Thus, E-SNRHT aims to broaden the reach of HIV testing to people who are reluctant to participate in risk partner recruitment. Network members recruited by a seed will also be asked to recruit additional people they know using the same education and recruitment instructions provided to seeds. All network members will be tested for HIV and provided with pre- and post-test counseling, all participants diagnosed with HIV will be referred to care, and all participants who test negative for HIV will be referred to 3-month follow-up HIV testing.
  Interventions: Behavioral: Expanded Social Network Recruitment to HIV Testing (E-SNRHT) Intervention
- Control Arm (No Intervention): The control arm consists of usual standard of care HIV testing and treatment at DoH clinics. In this arm, people newly diagnosed with HIV at clinics randomly assigned to the control condition will be recruited as control arm participants. They will be recruited and interviewed, and their HIV viral load will be measured. They will be encouraged to follow up with the clinic at which they were diagnosed for usual standard HIV care.

INTERVENTIONS:
Behavioral: Expanded Social Network Recruitment to HIV Testing (E-SNRHT) Intervention — The E-SNRHT intervention will recruit people newly diagnosed with HIV as "seeds," briefly remind them of HIV transmission risks and how HIV spreads through networks, and ask them to recruit people in their expanded social networks (i.e., anyone they know) who they think might benefit from being tested for HIV, regardless of whether or not they have engaged in any HIV risk behaviors together. By including expanded social networks, E-SNRHT aims to broaden the reach of HIV testing to people who are reluctant to participate in risk partner recruitment and/or to seek clinic testing. Network members recruited by a seed will also be asked to recruit additional people they know using the same education and recruitment instructions provided to seeds. All network members will be tested for HIV and provided with pre- and post-test counseling, all participants diagnosed with HIV will be referred to care, and all participants who test negative will be referred to 3-month follow-up HIV testing.
  Arms: E-SNRHT Intervention Arm

SUMMARY:
In South Africa's large generalized HIV epidemic, male-to-female transmission comprises a large proportion of transmission events, but men are much less likely to seek HIV testing, and disproportionately remain undiagnosed. HIV-related stigma is a key barrier to recruiting men to HIV testing in South Africa, as they report feeling blamed by their partners and communities for HIV transmission. This barrier must be addressed to increase testing among men and other testing-avoidant people in order to locate "hard-to-reach" undiagnosed cases and make progress towards 95-95-95 goals. Peer recruitment via social networks is an effective mechanism for promoting HIV testing, because people seek health information from peers, and peers influence health behavior norms within networks. However, standard risk network recruitment is limited in that: 1) recruiting one's own risk partners can trigger stigma and blame for HIV; and 2) it excludes people who have not engaged in HIV risk behavior recently and/or who no longer have contact with their risk partners. The Investigative Team for the present study developed an expanded social network recruitment to HIV testing (E-SNRHT) intervention to address these limitations and reduce stigma as a barrier to testing. E-SNRHT asks "seeds" (i.e., initial participants) who have been newly diagnosed with HIV (NDH) to recruit their expanded social network members (i.e., anyone they know) who they think could benefit from HIV testing or could have an undiagnosed HIV infection, tests these network members, and refers them to ART (if positive) or follow-up testing (if negative). By asking participants to recruit non-risk partners, E-SNRHT is designed to increase their comfort and likelihood of recruiting others, especially those who have avoided testing due to stigma. The Investigative Team's two previous pilot studies of E-SNRHT found that it recruits men to HIV testing at much higher rates than standard risk network recruitment; locates people with newly diagnosed HIV (PNDH; i.e., people with previously undiagnosed HIV infection) at a much higher rate per seed than standard risk network recruitment; and recruits people who have not tested in years, have never tested, and/or have not engaged in HIV risk behavior recently but have undiagnosed HIV infection. These pilot studies also found that E-SNRHT reduces HIV-related stigma and increases HIV-related social support among networks; and that 76% of E-SNRHT participants who were NDH started ART within 10 weeks. As participants recruit each other, their discussions help to normalize talking about HIV, thereby improving levels of stigma and support, which in turn should increase HIV service use and improve HIV care cascade outcomes. The present study will conduct a site-randomized trial of E-SNRHT, with 32 Department of Health clinics in KwaZulu-Natal, South Africa serving as sites. This study will compare E-SNRHT clinics to business-as-usual control clinics on: their rates of recruiting men to testing (Aim 1a) and locating PNDH (1b); participants' reports of HIV-related stigma and social support (Aim 2a); and treatment cascade outcomes (2b). Implementation science methods and qualitative methods will also be used to develop best practices (Aim 3) for future scale-up in South Africa and adaptation to other settings.

DETAILED DESCRIPTION:
Study Overview. The primary goal of the proposed study is to conduct a site-randomized trial (with Department of Health [DoH] clinics in the Msunduzi region of KwaZulu-Natal, South Africa as sites) to evaluate the efficacy of an expanded social network recruitment to HIV testing (E-SNRHT) intervention that is designed to extend the reach of HIV testing and care to groups and individuals that have been "hard-to-reach" for HIV testing, and to address HIV-related stigma as a barrier to HIV testing. Thirty-two participating DoH clinics will be randomly assigned to either the E-SNRHT intervention condition or to the control condition using urbanicity-stratified random assignment. People with newly-diagnosed HIV (PNDH) will then be recruited at participating clinics as "seeds" (i.e., initial study participants). After conducting brief education to remind them of HIV transmission risks and how HIV transmits through networks, seed participants in the intervention arm only (i.e., seeds recruited from an intervention condition-assigned clinic) will be asked to recruit members of their expanded social networks (e.g., friends, family members, acquaintances) who they think may be at risk of having undiagnosed HIV infection, or may otherwise benefit from HIV testing. All recruited network members will be tested for HIV, and will then be referred to additional HIV services: (i) those who test positive for HIV will be referred to antiretroviral treatment (ART) and offered support with appointment scheduling and navigating the clinic system, and (ii) those who test negative for HIV will be offered support to schedule follow-up HIV testing at 3 months and 6 months post baseline. This intervention not only aims (a) to increase rates of HIV testing and care among groups who test at low rates in this setting (specifically to men, who test in Msunduzi area clinics at much lower rates than women); and (b) to locate previously undiagnosed cases of HIV at higher rates than business as usual clinic testing; but also aims (c) to reduce HIV-related stigma and increase HIV-related social support through the process of peer recruitment, which will facilitate and normalize conversations about HIV and related services among peer networks. All participants will be interviewed and assessed at baseline, and will also be asked to complete 6-month follow-up interviews. A subset of 50 participants who are network members will also be asked to participate in in-depth qualitative interviews about their experiences being recruited to HIV testing by peers and recruiting their peers to HIV testing. Implementation data will also be collected based on the RE-AIM implementation science framework, in order to evaluate implementation success on key RE-AIM outcomes.

Recruitment Coupons. All recruitment of participants' network members in the intervention condition will occur via the distribution of recruitment coupons by participants. Coupons will contain unique, confidential alpha-numeric codes which will not contain any identifying information about the participant, but which will be used to link participants' social network members to them for analytic purposes. To protect participants' privacy, coupons will state only that the study is about "community health." Coupon design and language (and all study materials and procedures) will be reviewed and approved by UIC's and HSRC's IRBs and HSRC's Community Advisory Board (CAB) that HSRC maintains in the study locality, comprised of diverse, representative community stakeholders. The PIs will meet several times with the CAB during the recruitment period to report recruitment rates by site, to ensure there are no concerns with variation in recruitment being indicative of participants' discomfort with recruitment procedures at some sites.

Number and Characteristics of Participants to Be Enrolled. A planned total of 2,480 human subjects will be involved in the proposed research. Of these, 560 will be "seed" participants (i.e., original trial participants) who are newly-diagnosed with HIV (NDH), recruited from "business as usual" HIV testing at 32 Department of Health (DoH) clinics in the Msunduzi region of KwaZulu-Natal, South Africa. The remaining 1,920 participants will be the expanded social network members of intervention arm seeds, who will be recruited to the study by seed participants.

The 32 Department of Health clinics included in the study will include 10 clinics in urban areas, 10 clinics in suburban areas, and 12 clinics in rural areas. These 32 clinics will be randomly assigned to the expanded social network recruitment to HIV testing (E-SNRHT) intervention condition or to the control condition using urbanicity-stratified random assignment to ensure that conditions are balanced within each urbanicity type, before participant enrollment begins. Seed participants and the network members they recruit will therefore be enrolled into the study condition (intervention or control condition) already assigned to the clinic at which they (the seeds) were diagnosed with HIV and recruited to the study.

A planned 15 seeds from each of the 16 intervention clinics and 20 seeds from each of the 16 control clinics (240 intervention seeds + 320 control seeds = 560 total seeds) will be recruited. Seeds recruited from intervention condition clinics will be asked to recruit their expanded social network members to the study, and seeds recruited from control condition clinics will not. Specifically, seeds recruited from intervention clinics will be shown a diagram of how HIV spreads through a community and reminded of potential HIV transmission risk behaviors, and then asked to recruit anyone they know (e.g., friends, family members) who they think might be at risk of having undiagnosed HIV infection, or who they think might otherwise benefit from being tested for HIV, regardless of whether or not they have engaged in any HIV risk behaviors together. By including expanded social network members who participants perceive to be at risk of having undiagnosed HIV infection, this approach aims to broaden the reach of HIV testing to people who have previously been "hard-to-reach" for HIV testing.

Network member recruitment will follow a "two steps" algorithm for the E-SNRHT intervention arm, meaning that all participants who are recruited by intervention seeds (i.e., Step 1 network members) will also be asked to help the study recruit additional people they know who they think would benefit from HIV testing (i.e., Step 2 network members). If network members are not PNDH (i.e., people with undiagnosed HIV who are first diagnosed by the study team during the study), recruitment will end with Step 2 network members. However, a "2-steps from any PNDH" algorithm will also be used, such that if a Step 1 or Step 2 individual is found to be NDH, recruitment of people in his or her network will continue until two steps have been completed without recruiting another PNDH. This algorithm will maximize E-SNRHT's ability to locate PNDH and link them to care.

The Investigative Team's previous 2022-2023 pilot study of the intervention found an average network size of 6.5 network members for each seed. To account for the extension of network recruitment beyond Step 2 for networks that recruit PNDH (i.e., to account for the "2-steps from any PNDH" algorithm described above, which was not used in the pilot), total expected enrollment has been based on an average expected total network size of 8 network members per seed. The total approximate N of network members = 8 network members x 15 seeds x 16 sites = 1,920. The total anticipated sample is thus 2,480 (1,920 network members + 240 intervention seeds + 320 control seeds).

As stated above, participants will be recruited from clinics in the Msunduzi region. This region is comprised mostly of isiZulu- and English-speaking populations of Zulu heritage, but includes some areas with large English-speaking white and Indian populations. It is characterized by high HIV prevalence and incidence, high rates of unemployment, and low per capita income. Based on pilot data, up to 33% of network members are expected to be people living with HIV (15% PNDH [i.e., people with previously undiagnosed HIV infection who will be diagnosed during the study], plus up to 18% who were diagnosed with HIV before study participation, since participants are recruiting people they perceive to be at high risk for HIV but whose status they do not know).

Testing. At the time of the baseline interview, rapid HIV tests will be conducted for all network members. Before reviewing the results of the HIV test, pre-test counseling will be provided. After providing participants with their HIV test results, additional post-test counseling will also be provided. All participants who receive positive HIV test results will also receive a second, confirmatory HIV rapid test. All participants (including all seeds in both study arms) with diagnosed HIV infection will then be asked to provide a 5 milliliter (mL) blood sample for conducting a laboratory test of HIV viral load. Participants with diagnosed HIV infection will also be asked for 5 mL whole blood samples at the time of their 6-month follow-up interviews, for the purpose of measuring changes in viral load.

Referrals to Treatment or Additional HIV Testing. All participants who test positive for HIV will be referred to HIV treatment. After their interviews, E-SNRHT intervention arm participants who have been diagnosed with HIV (or were already aware that they were living with HIV) will be assisted by study referral staff in making clinic appointments. They will be given phone and email information to reach referral staff any time they need help in navigating the process of working with clinics to receive care. Approximately 2 months after their initial positive test, referral staff will contact them again to ask if they want additional help making follow-up appointments. All intervention arm participants who test negative for HIV at baseline will also be encouraged by study referral staff to schedule follow-up HIV testing appointments at a DoH clinic at 3-month intervals. All intervention arm participants will be assisted by study referral staff in making clinic appointments (for regular testing if they tested negative for HIV during the study, or for treatment if they have diagnosed HIV infection).

Baseline Quantitative Interviews. All participants will be interviewed about their sociodemographic characteristics, sexual and drug use behaviors during the last six months, previous use of HIV-related health services including antiretroviral therapy (ART - which is relevant since some network members may have long-diagnosed HIV infection), experiences of stigma and social support, and their perception of the level of HIV stigma in their communities. Audio computer-assisted structured interviewing (ACASI) will be u sed to ask questions about sensitive topics such as drug use and sexual behavior, such that participants will not have to answer these questions out loud.

Intervention arm participants who are asked to recruit network members (i.e., seeds and Step 1 network members) will be asked about the targeted members of their social networks who they will help recruit to the study. As described above, they will be asked to enumerate people in their expanded social networks (i.e., friends, family, peers, etc.) to recruit to the study who they believe might be at risk of having undiagnosed HIV infection, or would benefit from HIV testing. Participants asked to recruit others will be asked about the nature (i.e., type) and strength of their relationships to the network members they enumerate and plan to recruit, as well as about their basic descriptive characteristics like gender and approximate age. Their network members who enroll will also be asked about their relationship to the person who recruited them to the study.

All instruments to be used for the proposed study will be adapted from existing instruments that have been used for the Investigative Team's pilot studies of the E-SNRHT intervention in the Msunduzi area, and/or that have been validated for use with vulnerable populations. Any instrument that has not yet been used among the study population will be adapted for use among a predominately Zulu-background population, will be translated to isiZulu and back-translated to English by staff who are highly fluent in both languages (with translation and back-translation being completed by different staff members), and will be reviewed by the Community Advisory Board (CAB) prior to use in the proposed study.

Follow-up Quantitative Interviews. Participants will be asked to return to complete follow-up interviews approximately 6 months after their baseline interviews. For all participants, each follow-up interview will ask about sexual and drug use behaviors, interaction with all HIV-related health services since the last study interview (including ART uptake and adherence for participants with diagnosed HIV infection, and HIV regular testing for participants who tested negative during the study), and perceptions and experiences of stigma and social support. Additionally, participants' perceptions of intervention acceptability, appropriateness, and feasibility will be measured during the 6-month follow-up interview. Any stigmatizing or other negative experiences reported during or since participation in the study will be followed up. Detailed information will be gathered on the nature of all such reported experiences, and each one will be carefully evaluated to determine whether it should be categorized as an Adverse Event. All participants reporting any stigmatizing experiences will be given referrals to counseling at the time of their follow-up interviews, regardless of whether the reported stigma experience is related to study participation or is found to be an Adverse Event.

In-depth Qualitative Interviews. A subsample of 50 Step 1 network members (since all Step 1 network members both experienced being recruited and were asked to recruit others) will be selected with whom to conduct in-depth semi-structured interviews approximately 1-2 months after their baseline interviews, in order to ask them about their experiences being recruited to HIV testing by their peers and recruiting others to HIV testing. The initial in-depth interview guide will include the following topics: anticipated and experienced stigma and support, how recruiters chose the time and location to discuss HIV testing, participants' own reactions to being recruited and the reactions of others they tried to recruit, conversational ease or awkwardness, conversational content, and anticipated comfort with having future conversations about HIV with peers. Since this research is exploratory, additional topics may arise in early interviews that will be added to interview guides for subsequent participants.

Implementation Fidelity Data. To ensure protocol fidelity, fidelity checklist data will be collected to quantify and visualize how closely staff are adhering to implementation protocols, including: how frequently staff are delivering trainings within the targeted length of time, distributing study pamphlets correctly, referring study participants to correct follow-up services based on their HIV test results, contacting participants at the 3-month follow-up to schedule appointments, and quickly responding to participant requests for services. These data will be used to compute overall and staff-specific fidelity, defined as meeting 85% of intervention components. If staff fall below this threshold, the Investigators will re-train them to ensure they meet fidelity criteria.

Clinic Data On Service Uptake. Individual-level data will be collected from the 32 Department of Health (DoH) clinics participating in the proposed study at the time of follow-up data collection, on study participants' ART enrollment and initiation (for participants who have been diagnosed with HIV infection), and on HIV testing (for participants who tested negative for HIV at baseline). For participants who have obtained any of these services from the study-participating DoH clinics, data will be obtained on the date of initiation of ART and/or on the date of all HIV tests participants obtained during the study period. During the informed consent process, participants will be asked to indicate whether or not they consent to have the study obtain their HIV service access records from the DoH clinics. As an additional comparison to the outcomes of intervention participants, aggregate clinic-level data will also be obtained from the DoH clinics at both baseline and follow-up on their numbers and proportions of men and women who received standard of care HIV testing, on the proportions of HIV tests that resulted in new HIV diagnoses, and on the numbers and proportions of NDH clinic patients who initiated ART and/or achieved viral suppression during baseline and follow-up data collection periods. The DoH regularly computes and shares these aggregate clinic-level indicators with HSRC as part of a standing data sharing agreement, and the broader study team has permission to access these data during the study period.

Participant Locator Forms. All participants will be asked to complete a locator form at the time of their baseline interviews so that this information can be used to contact them to complete follow-up interviews. Participants will be informed during the consent process about this follow-up component and will be informed that study staff will contact them again before their 6-month follow-up interviews (and to possibly contact them about 1-2 months after their baseline interviews to ask them to participate in an in-depth qualitative interview). Locator forms will include the participants' own contact information, as well as information about other individuals who might be able to help locate the participant if the study team is unable to do so directly.

Outcomes to Be Compared between Study Arms to Evaluate Intervention Efficacy. Outcomes to be compared between intervention and control arms to evaluate the efficacy of the E-SNRHT intervention are: proportion of people tested in each study arm who are men; proportion of people tested in each study arm who are NDH; experiences and perceptions of HIV-related stigma; experiences and perceptions of HIV-related support; ART initiation; and HIV viral suppression.

ELIGIBILITY:
"Seeds" (i.e., initial participants in both study arms) will be recruited via referrals from clinics' standard of care HIV testing. To be eligible, seeds must have received a new HIV diagnosis from a study clinic in the last 2 months (i.e., they must be newly diagnosed with HIV infection [NDH]), and must have been given a study recruitment coupon by staff at one of these clinics. They will also be screened to ensure that they meet the following additional eligibility criteria: are ≥ 18 years old, are able to be interviewed in English or isiZulu (since over 95% of the population in the Msunduzi region speaks one or both of these languages), are able to give informed consent, and indicate that they reside in the Msunduzi region of KwaZulu-Natal, South Africa.

Seeds in the intervention arm (i.e., recruited from intervention condition-assigned clinics) will be asked to recruit their expanded social network members who they think would benefit from testing for HIV. Network members will be eligible to participate if they have a recruitment coupon given to them by a study participant (i.e., if they were recruited by an intervention arm participant); are ≥ 18 years old; able to be interviewed in English or isiZulu; able to give informed consent; and reside in the Msunduzi region.

Inclusion Criteria:

* Has study recruitment coupon (from clinic or from intervention arm participant)
* Is ≥ 18 years old
* Is able to be interviewed in English or isiZulu
* Is able to give informed consent
* Resides in the Msunduzi region

Exclusion Criteria:

* Does not have study recruitment coupon (from clinic or from intervention arm participant)
* Is < 18 years old
* Is not able to be interviewed in English or isiZulu
* Is not able to give informed consent
* Does not reside in the Msunduzi region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2480 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Rates of men recruited to HIV testing | Baseline
  Rates of men recruited to HIV testing will be computed at the clinic site level, using routine clinic testing data to calculate proportions of patients tested at control sites during the baseline study enrollment period who are men. At intervention sites, the proportion of all network-recruited participants from each site who are men will be calculated, to facilitate comparison of the E-SNRHT intervention with business as usual clinic testing procedures.
Rates of people newly-diagnosed with HIV by the intervention (i.e., people with previously-undiagnosed HIV infection) | Baseline
  People newly diagnosed with HIV by the intervention (PNDH) will be defined as participants who test positive for HIV, have no recorded previous positive HIV test, and indicate to clinic or study staff that they have never received a positive HIV test result before. Rates of PNDH will be computed at the clinic site level, using routine clinic testing data to calculate proportions of patients tested at control sites during the baseline study enrollment period who are newly diagnosed with HIV (NDH). At intervention sites, the proportion of all network-recruited participants from each site who are NDH will be calculated, to facilitate comparison of the E-SNRHT intervention with business as usual clinic testing procedures.
Individual-level experiences of HIV-related stigma | baseline and 6-month follow-up
  Participants' direct experiences of HIV-related stigma will be measured using questions adapted from the Investigators' previous study which ask participants whether they have experienced specific stigmatizing behaviors upon someone learning or thinking that they had HIV.
Individual-level enacted HIV-related stigma (measured using HIV Stigma Scale) | baseline and 6-month follow-up
  Participants' individual experiences of HIV-related stigma will be measured using the enacted stigma items from the HIV Stigma Scale.
Social experiences related to participation in the study | baseline and 6-month follow-up
  To monitor potential harm of the intervention, participants will be asked whether or not they have had any of a specific list of negative social experiences that they believe to be related to their participation in the study.
Community-level HIV-related stigma | baseline and 6-month follow-up
  Perceptions of the amount of HIV-related stigma present in participants' communities will be measured using 7 dichotomous items from a measure developed by the PI's previous research team. These items, adapted from the Perceived Stigma of HIV/AIDS: Public Views Scale, ask how likely respondents think people living with HIV are to experience a set of stigmatizing responses from members of their community.

SECONDARY OUTCOMES:
Individual-level experiences of HIV-related social support | baseline and 6-month follow-up
  Participants' direct experiences of HIV-related social support will be measured using a) questions adapted from the Investigators' previous study which ask participants whether they have experienced specific helping/ supportive behaviors upon someone learning or thinking that they had HIV.
Participant antiretroviral treatment (ART) initiation | 6-month follow-up
  At follow-up, participants who were NDH at baseline will be asked about their ART access and use. These self-report data will be triangulated with clinic reports on individuals' receipt of ART. (Explicit consent will be obtained for this, giving participants the option on consent forms to deny the study access to this information.) These data will be used to calculate the proportion of NDH participants from each site who started ART by six-month follow-up. Measuring these outcomes with individual-level data will address any threat to internal validity due to participants getting HIV treatment at multiple clinics during the follow-up period.
Clinic-level rates of antiretroviral treatment (ART) initiation | 6-month follow-up
  Clinic-level proportions of PNDH (diagnosed during the baseline data collection period) who started ART within six months of diagnosis will be measured using routinely-collected clinic-level data.
Participant HIV viral suppression | 6-month follow-up
  Results of viral load tests conducted at follow-up will be used to calculate the proportion of NDH participants from each clinic site who achieved viral suppression (<50 copies/mL). Measuring these outcomes with individual-level data will address any threat to internal validity due to participants getting HIV treatment at multiple clinics during the follow-up period.
Clinic-level HIV rates of viral suppression | 6-month follow-up
  Clinic-level data will be used to compute, for each clinic site, the proportion of patients who started ART (since the beginning of the study) who reached viral suppression (as defined by the South African DoH) by the time of 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie D. Williams, Ph.D., Principal Investigator — University of Illinois Chicago
Locations (1):
- Centre for Community-based Research, Human Sciences Research Council, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
In keeping with the goal of maximizing data sharing, the Investigators will deposit de-identified project data in openICPSR©. The de-identified data will be preserved as-is and available to data users at no cost for a minimum of ten years. openICPSR© requires that data users must be granted approval for access.
  All data will be completely de-identified to ensure participant confidentiality. Users of the public use data will be required to register with ICPSR and agree to its Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, by prohibiting attempts to identify study participants, and by requiring immediate reporting of attempts to identify study participants, and by requiring immediate reporting of any disclosure of study participant identity. Data users will also be required to agree not to share or redistribute any data downloads.
Supporting Information: Study Protocol
Time Frame: Within 12 months of the publication of the set of papers that address the main specific aims of this study, all data will be compiled in a standard statistical software and available for open access. The data will be available for a minimum of ten years.
Access Criteria: OpenICPSR© is a secure repository for storing and sharing social and behavioral science research data. To ensure confidentiality and to protect sensitive data, openICPSR© reviews all data to assess disclosure risk and to determine the level of access (open or restricted). Additionally, openICPSR© requires that data users must be granted approval for access, and in cases of restricted data, allows access only via controlled virtual labs. Users of the public use data will be required to register with ICPSR and agree to its Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, by prohibiting attempts to identify study participants, and by requiring immediate reporting of any disclosure of study participant identity. Data users will also be required to agree not to share or redistribute any data downloads.
URL: https://www.openicpsr.org/openicpsr/